CLINICAL TRIAL: NCT02627872
Title: Clinical & Systems Medicine Investigations of Smoking-related Chronic Obstructive Pulmonary Disease
Acronym: COSMIC
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: University of California, San Francisco (Other); Göteborg University (Other); University of Bergen (Other); University of Oulu (Other); Kyoto University (Other); Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Region Stockholm (Other Government); Vinnova (Other Government); Swedish Foundation for Strategic Research (Other); European Union (Other)
Responsible Party: Principal Investigator, Asa Wheelock, Associate professor, Karolinska Institutet
Other Study IDs: 2006/959-31/1
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis; Chronic Airways Obstruction; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage (BAL) cells, BAL fluid, bronchial biopsies, airway epithelial brushings, serum, plasma, and blood cells have been collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- COPD patients (GOLD I-II): Participants with mild-to-moderate COPD (GOLD I-II)
- Smoker Control Group: Actively smoking participants with normal lung function (do not have COPD)
- Healthy Never-smoker Control Group: Healthy participants that never have smoked

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is an increasing global health problem, which primarily increases among the female population. The purpose of this study is to perform in-depth clinical and molecular characterizations of early stage COPD patients, as well as healthy never-smoker and at-risk smoking control populations to identify molecularly related subgroups patients, including gender-related sub-phenotypes of COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an umbrella diagnosis defined by obstructive lung function impairments, and is likely to be caused by a multitude of etiologies including environmental exposures, genetic predispositions and developmental factors. Due to the heterogeneity of the disease, molecular and mechanistic sub-phenotyping of COPD represents an essential step to facilitate the development of relevant diagnostic and treatment options for this constantly growing patient group. In the Karolinska COSMIC study, the investigators are investigating molecular sub-phenotypes of smoking-induced COPD. A particular focus relates to recent epidemiological indications of gender differences in both incidence and severity of disease, with post-menopausal women being at greatest risk. The study encompasses profiling of mRNA, miRNA, proteomes, metabolomes and lipid mediators of from multiple lung compartments (airway epithelium, alveolar macrophages, exosomes, and bronchoalveolar exudates) using a range of 'omics platforms, in combination with extensive clinical phenotyping of early stage COPD patients, never-smokers, and smokers with normal lung function from both genders. The primary objective of the study is to identify molecular sub-phenotypes of patients with COPD, specifically by correlating clinical phenotypes multi-molecular 'omics profiling from multiple lung compartments of early stage COPD patients compared to healthy and at-risk control populations. Secondary goals involve identification of subsets of prognostic/diagnostic biomarkers for classification of the defined subgroups, as well as relevant pharmaceutical targets.

ELIGIBILITY:
Inclusion Criteria:

* For smokers, at least 10 pack-years of cigarette smoking
* For smokers, at least 10 cigarettes/day the past 6 months before study entry Spirometry that meets stage I-II of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) stages (postbronchodilator forced expiratory volume in 1 second (FEV1) of 50%-100% of predicted level and FEV1/forced vital capacity [FEV1/FVC] less than 0.7) or normal (postbronchodilator FEV1 greater than 80% of predicted level and forced expiratory volume in 1 second/forced vital capacity [FEV1/FVC] greater than 0.7)

Exclusion Criteria:

* Other lung diseases
* Atopy (defined as positive specific IgE test)
* Asthma
* Received antibiotics for a COPD exacerbation in the 3 months prior to study entry
* Treatment with oral or inhaled glucocorticoids within past 3 months prior to study entry
* Significant ischaemic heart disease or arrhythmia

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from all groups are recruited from the general population through advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2021-12 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | Measured at baseline and up to 10 year follow-up
Emphysema, as shown on chest CT scan | Measured at baseline and up to 10 year follow-up
Airway wall thickness on chest CT scan | Measured at baseline and up to 10 year follow-up
COPD status (COPD participants versus control group participants) | Measured at baseline and up to 10 year follow-up
Molecular gender differences | Measured at baseline
  Molecular levels investigated: mRNA, miRNA, proteome, metabolome, lipidome

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet/Karolinska University Hospital Solna, Stockholm, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The deidentified clinical phenotype data has been disseminated through peer reviewed publication

REFERENCES:
- [Background] Sandberg A, Skold CM, Grunewald J, Eklund A, Wheelock AM. Assessing recent smoking status by measuring exhaled carbon monoxide levels. PLoS One. 2011;6(12):e28864. doi: 10.1371/journal.pone.0028864. Epub 2011 Dec 16. PMID 22194931
- [Result] Forsslund H, Mikko M, Karimi R, Grunewald J, Wheelock AM, Wahlstrom J, Skold CM. Distribution of T-cell subsets in BAL fluid of patients with mild to moderate COPD depends on current smoking status and not airway obstruction. Chest. 2014 Apr;145(4):711-722. doi: 10.1378/chest.13-0873. PMID 24264182
- [Result] Karimi R, Tornling G, Forsslund H, Mikko M, Wheelock A, Nyren S, Skold CM. Lung density on high resolution computer tomography (HRCT) reflects degree of inflammation in smokers. Respir Res. 2014 Feb 24;15(1):23. doi: 10.1186/1465-9921-15-23. PMID 24564813
- [Result] Kohler M, Sandberg A, Kjellqvist S, Thomas A, Karimi R, Nyren S, Eklund A, Thevis M, Skold CM, Wheelock AM. Gender differences in the bronchoalveolar lavage cell proteome of patients with chronic obstructive pulmonary disease. J Allergy Clin Immunol. 2013 Mar;131(3):743-51. doi: 10.1016/j.jaci.2012.09.024. Epub 2012 Nov 10. PMID 23146379
- [Result] Mikko M, Forsslund H, Cui L, Grunewald J, Wheelock AM, Wahlstrom J, Skold CM. Increased intraepithelial (CD103+) CD8+ T cells in the airways of smokers with and without chronic obstructive pulmonary disease. Immunobiology. 2013 Feb;218(2):225-31. doi: 10.1016/j.imbio.2012.04.012. Epub 2012 May 4. PMID 22652413
- [Result] Balgoma D, Yang M, Sjodin M, Snowden S, Karimi R, Levanen B, Merikallio H, Kaarteenaho R, Palmberg L, Larsson K, Erle DJ, Dahlen SE, Dahlen B, Skold CM, Wheelock AM, Wheelock CE. Linoleic acid-derived lipid mediators increase in a female-dominated subphenotype of COPD. Eur Respir J. 2016 Jun;47(6):1645-56. doi: 10.1183/13993003.01080-2015. Epub 2016 Mar 10. PMID 26965288
- [Result] Forsslund H, Yang M, Mikko M, Karimi R, Nyren S, Engvall B, Grunewald J, Merikallio H, Kaarteenaho R, Wahlstrom J, Wheelock AM, Skold CM. Gender differences in the T-cell profiles of the airways in COPD patients associated with clinical phenotypes. Int J Chron Obstruct Pulmon Dis. 2016 Dec 20;12:35-48. doi: 10.2147/COPD.S113625. eCollection 2017. PMID 28053515
- [Result] Karimi R, Tornling G, Forsslund H, Mikko M, Wheelock AM, Nyren S, Skold CM. Differences in regional air trapping in current smokers with normal spirometry. Eur Respir J. 2017 Jan 25;49(1):1600345. doi: 10.1183/13993003.00345-2016. Print 2017 Jan. PMID 28122862
- [Result] Naz S, Kolmert J, Yang M, Reinke SN, Kamleh MA, Snowden S, Heyder T, Levanen B, Erle DJ, Skold CM, Wheelock AM, Wheelock CE. Metabolomics analysis identifies sex-associated metabotypes of oxidative stress and the autotaxin-lysoPA axis in COPD. Eur Respir J. 2017 Jun 22;49(6):1602322. doi: 10.1183/13993003.02322-2016. Print 2017 Jun. PMID 28642310
- [Result] Li CX, Wheelock CE, Skold CM, Wheelock AM. Integration of multi-omics datasets enables molecular classification of COPD. Eur Respir J. 2018 May 10;51(5):1701930. doi: 10.1183/13993003.01930-2017. Print 2018 May. PMID 29545283
- [Result] Naz S, Bhat M, Stahl S, Forsslund H, Skold CM, Wheelock AM, Wheelock CE. Dysregulation of the Tryptophan Pathway Evidences Gender Differences in COPD. Metabolites. 2019 Oct 1;9(10):212. doi: 10.3390/metabo9100212. PMID 31581603
- [Result] Fuchs D, Hamberg M, Skold CM, Wheelock AM, Wheelock CE. An LC-MS/MS workflow to characterize 16 regio- and stereoisomeric trihydroxyoctadecenoic acids. J Lipid Res. 2018 Oct;59(10):2025-2033. doi: 10.1194/jlr.D087429. Epub 2018 Jul 31. PMID 30065010
- [Result] Che KF, Tufvesson E, Tengvall S, Lappi-Blanco E, Kaarteenaho R, Levanen B, Ekberg M, Brauner A, Wheelock AM, Bjermer L, Skold CM, Linden A. The neutrophil-mobilizing cytokine interleukin-26 in the airways of long-term tobacco smokers. Clin Sci (Lond). 2018 May 20;132(9):959-983. doi: 10.1042/CS20180057. Print 2018 May 23. PMID 29780024
- [Result] Che KF, Kaarteenaho R, Lappi-Blanco E, Levanen B, Sun J, Wheelock A, Palmberg L, Skold CM, Linden A. Interleukin-26 Production in Human Primary Bronchial Epithelial Cells in Response to Viral Stimulation: Modulation by Th17 cytokines. Mol Med. 2017 Oct;23:247-257. doi: 10.2119/molmed.2016.00064. Epub 2017 Aug 29. PMID 28853490
- [Result] Merikallio H, Kaarteenaho R, Linden S, Padra M, Karimi R, Li CX, Lappi-Blanco E, Wheelock AM, Skold MC. Smoking-associated increase in mucins 1 and 4 in human airways. Respir Res. 2020 Sep 18;21(1):239. doi: 10.1186/s12931-020-01498-7. PMID 32948202
- [Result] Yang M, Kohler M, Heyder T, Forsslund H, Garberg HK, Karimi R, Grunewald J, Berven FS, Magnus Skold C, Wheelock AM. Long-term smoking alters abundance of over half of the proteome in bronchoalveolar lavage cell in smokers with normal spirometry, with effects on molecular pathways associated with COPD. Respir Res. 2018 Mar 8;19(1):40. doi: 10.1186/s12931-017-0695-6. PMID 29514648
- [Result] Yang M, Kohler M, Heyder T, Forsslund H, Garberg HK, Karimi R, Grunewald J, Berven FS, Nyren S, Magnus Skold C, Wheelock AM. Proteomic profiling of lung immune cells reveals dysregulation of phagocytotic pathways in female-dominated molecular COPD phenotype. Respir Res. 2018 Mar 8;19(1):39. doi: 10.1186/s12931-017-0699-2. PMID 29514663